CLINICAL TRIAL: NCT02236143
Title: Ultrahigh Field Body MR Imaging
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1212M24883
Record Dates: First submitted 2013-03-13; First posted 2014-09-10 (Estimated); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Structure and Function of MRI
Keywords: Healthy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MRI: Subjects undergoing MRI

SUMMARY:
The primary objective of this study is to develop new ways to acquire MRI data and/or new ways to analyze the acquired data.

DETAILED DESCRIPTION:
The acquired data will be used to investigate the structure and function of the body. In addition the developmental aspect of this study, certain information may be used to obtain normal values for healthy adult structural and functional information. This information would be valuable if and when the developed methods are incorporated into future clinical studies involving patient populations which would be recruited under separate protocols. Our hypotheses is that imaging and spectroscopy methods can be developed to a level where the increased sensitivity and resolution of 7 Tesla (7T) MRI will improve the non-invasive studies of the human body.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteer over the age of 18

Exclusion Criteria:

* Exclusion criteria include those associated with the use of MR as the imaging modality. The specific set of exclusion criteria for a given study will depend on the specific study to be performed which will be made clear on initial contact and during consent. In addition, other medical conditions deemed by the PI or associates to make the patient ineligible for protocol procedures may also arise.
* Exclusion criteria will be assessed during a safety screening interview and during final consent. A questionnaire will be provided regarding general health and exclusion/inclusion criteria. The investigator doing the interview will determine if any of the exclusion criteria apply. Subjects will be asked:

  1. To describe any previous surgeries to help subjects and study staff open a dialogue as to any possible contraindications listed in the yes/no section below.
  2. If they are claustrophobic and to rate the severity.
  3. If they wear hearing aids and if they can be removed for the scan.
  4. If they have a transdermal delivery system, and if yes where is it located and if it can be removed for the study.
  5. If they wear colored contact lenses and, if yes, can they be removed for the study.
  6. To provide a list of medications, dosages and time of last dose for medicines taken regularly.
  7. To identify if they have any pre-existing medical conditions including Hypertension, Hypotension, Diabetes, Cardiovascular Disease and Fever.
  8. To identify if they ever had an operation.
  9. To indicate if they have ever been injured by a metallic foreign body which was never removed.
  10. If they wear braces and/or if they have removable bridgework, false teeth or a permanent retainer.
  11. If they have any tattoos, non-removable body piercings or hair extensions.
  12. If they are currently using/wearing an IUD or diaphragm.
  13. If they have any reason to believe they are pregnant. (If the subjects are unsure about their pregnancy status, test kits will be available to subjects).
* In addition, a set of yes/no questions will be asked in the screening form for the patient to confirm or deny the presence of items that may be hazardous to their safety and/or some interfere with the MRI examination, including:

No Cardiac pacemaker

No Implanted cardiac defibrillator

No Carotid artery vascular clamp

No Intravascular stents, filters, or coils

No Aortic clip

No Internal pacing wires

No Vascular access port and/or catheter

No Swan-Ganz catheter

No Shunt (spinal or intraventricular)

No Aneurysm clip(s)

No Neurostimulator

No Electrodes (on body, head, or brain)

No Heart valve prosthesis

No Any type of prosthesis (eye, penile, etc.)

No Artificial limb or joint replacement

No Bone growth/fusion stimulator

No Bone/joint pin, screw, nail, wire, plate

No Metal rods in bones

No Harrington rods (spine)

No Metal or wire mesh implants

No Wire sutures or surgical staples

No Insulin pump or infusion device

No Any metal fragments (i.e. metal shop)

No Any implant held in place by a magnet

No Cochlear, otologic, or ear implant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male or females over the age of 18, recruiting by invitation only.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-02-01 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Structure and Function of MRI | Baseline
  Validate MRI measurement

CONTACTS AND LOCATIONS:
Overall Officials: Greg Meztger, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota CMRR, Minneapolis, Minnesota, United States